CLINICAL TRIAL: NCT03542058
Title: Detecting and Treating Subclinical Anthracycline Therapy Related Cardiac Dysfunction in Low Income Country
Acronym: SATRACD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Makerere University (Other)
Collaborators: University of Cape Town (Other); Uganda Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cardio-oncology study
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Chemotherapy Related Cardiac Dysfunction
MeSH Terms: interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Study participants will receive carvedilol for a period of 6 month. The initial dosage of carvedilol will be 3.125mg twice daily. Dosage will be titrated up two weekly until the maximum tolerable dose or ceiling dose of 25mg twice daily has been reached.
  Interventions: Drug: Carvedilol
- Control Group (No Intervention): Study participant will not receive any cardiac medication, apart from standard cancer care.

INTERVENTIONS:
Drug: Carvedilol — Participants who are randomized to treatment group will receive carvedilol for a period of 6 month.
  Other Names: Carvedilol Denk
  Arms: Treatment Group

SUMMARY:
The objective of this research is to describe the burden of subclinical anthracycline therapy related cardiac dysfunction( ATRCD) by applying international guideline on Uganda cancer patient and to evaluate the significance of treating subclinical ATRCD with carvedilol.

DETAILED DESCRIPTION:
Specific objectives:

1. To determine the incidence of subclinical ATRCD among cancer patient who receives Anthracycline therapy.
2. To compare the changes of GLS value between hypertension and non hypertension cancer patient at the competition of the anthracycline therapy.
3. To determine the correlation of conventional echocardiograghy(ECHO) parameters (MAPSE, S') with GLS, and their ability to diagnose or rule out subclinical ATRCD.
4. To determine the correlation of oxidative stress with cardiac function(GLS value) in patients who receives Anthracycline therapy
5. To describe the cardioprotective effect of carvedilol in patients with subclinical ATRCD.

METHODS This is going to be two prospective cohort study (cohort 1 and 2) followed by a randomized controlled trial (cohort 3).

To achieve objective 1 ,3 and 4, Cohort 1 will consecutively recruit 300 adult non hypertension cancer patients who are going to receive anthracycline therapy.

To achieve objective 2, Cohort 2 will consecutively recruit 53 adult hypertension cancer patients (group H) and 106 non hypertension controls (group N) who are going to receive anthracycline therapy. Controls will be recruited from cohort 1 by systemic sampling( Choosing the 2nd patients as they are enrolled in cohort 1).

Patient's demographic data, cancer diagnosis, dosage of anthracyclin, past medical history, symptoms, physical examinations, ECG, ECHO and laboratory data will be collected at the baseline. Patient follow up will be performed at the completion of the chemo therapy, and 6month thereafter. Data of symptoms, physical examinations, ECG, ECHO and blood test will be collected at each visit. The end point will be the development of subclinical ATRCD.

To achieve objective 5, patients in Cohort 1, who are diagnosed with Subclinical ATRCD will be recruited into cohort 3 and being randomized into group T(carvedilol treatment group) and group C( control, none treatment group).Systemic randomization will be used in Cohort 3: ever second eligible patient will be recruited in group C. Patients in cohort 3 will be followed up for 6month.

ELIGIBILITY:
Inclusion Criteria:

1. Age between and include 18 and 50 years.
2. Newly diagnosed cancer patients who develop subclinical ATRCD during cardiac follow up.

Exclusion Criteria:

1. Patient who has been taking carvedilol prior to the study
2. Patient who self report to be allergic to carvedilol
3. Systolic blood pressure < 90mmHg
4. Heart Rate < 50 beat per minute
5. Patient who is asthmatic or has chronic obstructive lung disease
6. Pregnant woman

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Cardiac function | 6 months
  This will be measured by mean GLS(Global Longitudinal strain) value.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sliwa, PhD, Study Chair — Hatter Institute for Cardiovascular Disease in Africa; Feriel Azibani, PhD, Study Director — Hatter Institute for Cardiovascular Disease in Africa

IPD SHARING:
Plan to Share IPD: Undecided